CLINICAL TRIAL: NCT02853591
Title: A Randomized-Controlled Trial of Conventional Pneumoinsufflation and Pressure-Barrier Insufflation at High and Low Pressures in Gynecologic Surgery
Brief Title: Comparison of Pneumoinsufflation Modes and Pressure Settings in Gynecology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: CONMED Corporation (Industry)
Responsible Party: Principal Investigator, Pamela Frazzini Padilla, Clinical Fellow, The Cleveland Clinic
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: FLA 16-056
Record Dates: First submitted 2016-07-26; First posted 2016-08-03 (Estimated); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Pain; Pneumoperitoneum; Inflammation; Quality of Life
Keywords: laparoscopy; hysterectomy
MeSH Terms: conditions — Pain; Pneumoperitoneum; Inflammation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Standard High Pressure (15mmHg) (Active Comparator): Pneumoinsufflator mode and setting: standard at 15mmHg
  Interventions: Procedure: Pneumoinsufflator mode and setting
- AirSeal High Pressure (15mmHg) (Experimental): Pneumoinsufflator mode and setting: pressure-barrier at 15mmHg
  Interventions: Procedure: Pneumoinsufflator mode and setting
- Standard Low Pressure (9mmHg) (Experimental): Pneumoinsufflator mode and setting: standard at 9mmHg
  Interventions: Procedure: Pneumoinsufflator mode and setting
- AirSeal Low Pressure (9mmHg) (Experimental): Pneumoinsufflator mode and setting: pressure-barrier at 9 mmHg
  Interventions: Procedure: Pneumoinsufflator mode and setting

INTERVENTIONS:
Procedure: Pneumoinsufflator mode and setting — Patients undergoing total laparoscopic hysterectomy will be randomized to pneumoperitoneum creation by one of two modes (standard or pressure-barrier) at one of two set pressures (15mmHg or 9mmHg) for a four-armed factorial designed study.
  Other Names: Intra-abdominal pressure

SUMMARY:
This study seeks to evaluate post-operative patient pain and quality of life, and intra-operative hemodynamic status and changes in inflammatory markers, with use of a pressure-barrier insufflator and conventional insufflator at high and low pneumoperitoneum pressure settings.

DETAILED DESCRIPTION:
This is a randomized-controlled double-blinded trial examining outcomes from total laparoscopic hysterectomies performed under low and high pressure pneumoperitoneum with either a novel pressure-barrier insufflator (AirSeal®) or conventional insufflator. All patients scheduled for total laparoscopic hysterectomy (without robotic-assistance) will be screened for eligibility in the study. If eligible, a standard informed consent process will ensue.

All research activities will commence on the day of surgery, in the pre-operative preparation area. Enrolled subjects will undergo standard registration and pre-operative preparation by the staff preoperative nurse, including placement of intravenous access line and administration of standard pre-operative intravenous medications (typically ondansetron, dexamethasone, and ketorolac). While in the pre-operative area, and prior to any sedative drug administration by anesthesia, the patient will complete an 11-point Numeric Rating Scale (NRS) for baseline pain, as well as a baseline 18-question quality of life survey with the Abdominal Surgery Impact Scale (ASIS). Both study instruments will be self-administered by the patients and collected by the research team. A baseline blood collection will be performed in the pre-operative area by the research team assistant and sent for inflammatory markers.

The subject will be moved to the operating room and the anesthesia team will apply the pads for use with the Cheetah Non-Invasive Cardiac Output Monitoring (NICOM) system, in addition to other standard anesthesia monitoring equipment. The Cheetah NICOM will be activated for baseline measurements prior to anesthesia induction. Induction, intubation, and anesthesia administration will be performed according to standard practice by a dedicated group of anesthesia providers. A second set of hemodynamic measurements from the Cheetah NICOM will be measured after intubation, prior to pneumoperitoneum. A select group of anesthesia providers familiar with the protocol will administer anesthesia using non-depolarizing muscle relaxants continuously adjusted to be no less than one twitch during pneumoperitoneum.

Prior to any incision, preoperative prophylactic antibiotics and surgical sterile preparation will be performed per usual technique. Bilateral upper extremities will be placed in a tucked position, and no shoulder pads will be used in any case. An 18g peripheral IV (ideally antecubital) will be placed to allow intra-operative blood draws. This may be placed before or after anesthesia induction, but prior to arm tucking.

Randomization will occur after the patient is anesthetized, but prior to surgical start time to allow proper equipment to be opened on the surgical field without waste. Randomization will be into one of four groups with equal allocation to each (1:1:1:1 ratio):

1. Conventional insufflation at 15mmHg intra-abdominal pressure. (Group 1)
2. Conventional insufflation at 9mmHg intra-abdominal pressure (Group 2)
3. AirSeal® insufflation at 15mmHg intra-abdominal pressure (Group 3)
4. AirSeal® insufflation at 9mmHg intra-abdominal pressure (Group 4) If randomized to an AirSeal® group, the tri-lumen filtered tube set and dedicated access trocar will be opened and placed on the surgical field. If randomized to the conventional insufflation group, conventional insufflation tubing with an additional conventional trocar will be opened and placed on the surgical field. The patient will remain blinded to randomization throughout the study, as will the research team assistant responsible for blood draws and administration of NRS and ASIS questionnaires.

Laparoscopic entry will typically be obtained by optical trocar in the periumbilical region, but placement may be modified at the surgeon's discretion. Initial pneumoperitoneum will be established through this trocar to a pressure of 15mmHg for all groups. Pressure will remain at this setting during Trendelenburg positioning and placement of other necessary laparoscopic trocars. Data will be recorded for the third time from the Cheetah NICOM at this point. Once all trocars are inserted, the AirSeal® system will be activated if necessary based on group randomization, and pressure will be decreased to 9mmHg if indicated based on randomization. Additional recordings of data from the Cheetah NICOM will occur 10 minutes and 30 minutes after pressure decrease, and the surgery will proceed according to the surgeon's preferred technique. Any surgeon-directed modifications of intra-abdominal pressure at any time for surgery completion and/or patient safety will be recorded.

Thirty minutes after pneumoperitoneum is established, the research team assistant will perform the second blood draw for inflammatory markers. The surgery will be completed per typical fashion, and total operative time and estimated blood loss will be recorded. A final Cheetah NICOM recording will be made 5 minutes after deflation of pneumoperitoneum.

The patient will emerge from anesthesia under their usual monitoring and be transferred to the post-anesthesia care unit (PACU) when meeting appropriate routine criteria. A staff PACU nurse will care for the subject in the PACU and administer pain medications as necessary and/or per patient request. All pain medication administration in the hospital will be recorded in the Epic electronic health record (EHR). The amount of each patient's narcotic administration will be recorded from the EHR and documented in study files. The staff PACU nurse will be blinded to subject group allocation.

The research team assistant will administer a NRS pain survey to the patient two hours post-operatively and inquire regarding presence of shoulder pain. The third blood draw will also occur at this timepoint by the research team assistant. All patients will undergo planned same-day discharge to home. If unable to be discharged, they will stay overnight in the hospital with documented rationale.

On the day after surgery, the subject will be contacted by the research team assistant who will administer a NRS pain survey by telephone (or in person if still in hospital) and ask patient to report number of narcotic pain pills used since discharge and dosage of each. Presence of shoulder pain will again be asked. If patient is still in the hospital, narcotic usage will be collected from the EHR.

Per standard routine, the patients will be asked to return to clinic two weeks post-operatively for evaluation and examination. The 18-question ASIS will be administered at this visit by the blinded research team assistant. If the patient cannot complete the "two-week visit" within 1-3 weeks after surgery, the research team assistant will administer the ASIS by telephone. The patient will exit the study after this visit. Blinding of the patient will be broken after administration of the ASIS, as it is standard practice to provide the patient with a copy of the operative report during this visit, which will describe the pneumoperitoneum settings used during their case.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet the following inclusion criteria to be eligible for the study.

  1. Understand and voluntarily sign an informed consent form.
  2. Female gender ages 18-65
  3. Scheduled for total laparoscopic hysterectomy for benign indications with or without oophorectomy (standard of care involves bilateral salpingectomy).

Exclusion Criteria:

* Meeting any of the following exclusion criteria will make the subject ineligible for the study.

  1. Anticipated removal of uterus through any route except vagina (transvaginal morcellation is acceptable)
  2. Planned concomitant procedures including but not limited to resection of deep endometriosis, plastic surgery procedures, or bowel resection.
  3. Daily narcotic pain medication use for greater than 30 days leading into surgery
  4. Use of da Vinci® robot surgical assistance

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-10; Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Pain score | 2 hours post-surgery
  Numerical rating scale

SECONDARY OUTCOMES:
Pain score on a NRS | 1 day post-surgery
  Numerical rating scale
Narcotic usage | 2 hours and 1 day post-surgery
  Morphine equivalents
Heart rate | Intra-operative (1. prior to anesthesia induction; 2. after induction prior to incision; 3. with pneumoperitoneum prior to Trendelenburg; 4. 10 minutes after trendelenburg; 5. 30 minutes after trendelenburg; 6. 5 minutes after pneumoperitoneum release
  beats per minute
Mean arterial pressure | Intra-operative (1. prior to anesthesia induction; 2. after induction prior to incision; 3. with pneumoperitoneum prior to Trendelenburg; 4. 10 minutes after trendelenburg; 5. 30 minutes after trendelenburg; 6. 5 minutes after pneumoperitoneum release
  mmHg
Total peripheral resistance | Intra-operative (1. prior to anesthesia induction; 2. after induction prior to incision; 3. with pneumoperitoneum prior to Trendelenburg; 4. 10 minutes after trendelenburg; 5. 30 minutes after trendelenburg; 6. 5 minutes after pneumoperitoneum release
  (mmHg*min)/mL
Oxygen saturation | Intra-operative (1. prior to anesthesia induction; 2. after induction prior to incision; 3. with pneumoperitoneum prior to Trendelenburg; 4. 10 minutes after trendelenburg; 5. 30 minutes after trendelenburg; 6. 5 minutes after pneumoperitoneum release
  oxygen saturation percent
Respiratory rate | Intra-operative (1. prior to anesthesia induction; 2. after induction prior to incision; 3. with pneumoperitoneum prior to Trendelenburg; 4. 10 minutes after trendelenburg; 5. 30 minutes after trendelenburg; 6. 5 minutes after pneumoperitoneum release
  breaths per minute
Tidal volume | Intra-operative (1. prior to anesthesia induction; 2. after induction prior to incision; 3. with pneumoperitoneum prior to Trendelenburg; 4. 10 minutes after trendelenburg; 5. 30 minutes after trendelenburg; 6. 5 minutes after pneumoperitoneum release
  liters
End tidal carbon dioxide | Intra-operative (1. prior to anesthesia induction; 2. after induction prior to incision; 3. with pneumoperitoneum prior to Trendelenburg; 4. 10 minutes after trendelenburg; 5. 30 minutes after trendelenburg; 6. 5 minutes after pneumoperitoneum release
  mmHg
Peak inspiratory pressure | Intra-operative (1. prior to anesthesia induction; 2. after induction prior to incision; 3. with pneumoperitoneum prior to Trendelenburg; 4. 10 minutes after trendelenburg; 5. 30 minutes after trendelenburg; 6. 5 minutes after pneumoperitoneum release
  mmHg
Stroke volume | Intra-operative (1. prior to anesthesia induction; 2. after induction prior to incision; 3. with pneumoperitoneum prior to Trendelenburg; 4. 10 minutes after trendelenburg; 5. 30 minutes after trendelenburg; 6. 5 minutes after pneumoperitoneum release
  mL
Stroke volume index | Intra-operative (1. prior to anesthesia induction; 2. after induction prior to incision; 3. with pneumoperitoneum prior to Trendelenburg; 4. 10 minutes after trendelenburg; 5. 30 minutes after trendelenburg; 6. 5 minutes after pneumoperitoneum release
  mL/beat/m^2
Stroke volume variation | Intra-operative (1. prior to anesthesia induction; 2. after induction prior to incision; 3. with pneumoperitoneum prior to Trendelenburg; 4. 10 minutes after trendelenburg; 5. 30 minutes after trendelenburg; 6. 5 minutes after pneumoperitoneum release
  stroke volume variation percent
Cardiac output | Intra-operative (1. prior to anesthesia induction; 2. after induction prior to incision; 3. with pneumoperitoneum prior to Trendelenburg; 4. 10 minutes after trendelenburg; 5. 30 minutes after trendelenburg; 6. 5 minutes after pneumoperitoneum release
  L/min
Cardiac index | Intra-operative (1. prior to anesthesia induction; 2. after induction prior to incision; 3. with pneumoperitoneum prior to Trendelenburg; 4. 10 minutes after trendelenburg; 5. 30 minutes after trendelenburg; 6. 5 minutes after pneumoperitoneum release
  L/min/m^2
Interleukin-6 (plasma) | Baseline (pre-anesthesia), intra-operative (30 minutes after Trendelenburg), 2 hours post-surgery
  pg/mL
C-reactive protein (plasma) | Baseline (pre-anesthesia), intra-operative (30 minutes after Trendelenburg), 2 hours post-surgery
  mg/dL
Tumor necrosis factor-alpha (plasma) | Baseline (pre-anesthesia), intra-operative (30 minutes after Trendelenburg), 2 hours post-surgery
  pg/mL
Epinephrine | Baseline (pre-anesthesia), intra-operative (30 minutes after Trendelenburg), 2 hours post-surgery
  pg/mL
Norepinephrine | Baseline (pre-anesthesia), intra-operative (30 minutes after Trendelenburg), 2 hours post-surgery
  pg/mL
Quality of life score based on the abdominal surgery impact scale | 2 weeks post-surgery
  Abdominal surgery impact scale
Conversion of low pneumoperitoneum to high pneumoperitoneum | Intra-operative (procedure start to finish)
  Number of subjects
Loss of pneumoperitoneum | Intra-operative (procedure start to finish)
  number of events
Total complications | Within first 30 days after surgery
  Vascular/bladder/ureter/intestinal injuries, blood transfusion, venous thromboembolism
Operative time | Intra-operative (procedure start to finish)
  minutes
Estimated blood loss | Intra-operative (procedure start to finish)
  mL

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Zimberg, MD, Principal Investigator — Cleveland Clinic Florida; Pamela Frazzini Padilla, MD, Principal Investigator — Cleveland Clinic Florida
Locations (1):
- Cleveland Clinic Florida, Weston, Florida, United States

IPD SHARING:
Plan to Share IPD: No